CLINICAL TRIAL: NCT06944821
Title: Effect of in Situ Simulation on Quality of Work Life and Multiprofessional Team Effectiveness in the Intensive Care Unit
Acronym: EFFIQUASS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RECHMPL24_0497
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Quality of Work Life; Burn-out; Simulation
Keywords: In-situ simulation; Intensive care; Stress; Quality of working life; Quality of care; Performance; Caregivers; Teamwork
MeSH Terms: conditions — Burnout, Psychological | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-situ stimulation (Experimental)
  Interventions: Procedure: In-situ simulation; Other: Role-playing using a simulation scenario; Other: Questionnaires
- Control (Other)
  Interventions: Other: Role-playing using a simulation scenario; Other: Questionnaires

INTERVENTIONS:
Procedure: In-situ simulation — Each simulation session takes place over one day, with 4 scenarios recreating life-threatening emergency situations (cardiorespiratory arrest, hemorrhagic shock, etc.). Each scenario is designed to meet specific pedagogical objectives, which will be debriefed by simulation trainers: crisis resource management (communication, alerting, etc.) or organization of multi-professional teamwork
  Arms: In-situ stimulation
Other: Role-playing using a simulation scenario — Team performance in critical situations, assessed during a simulation scenario for all participants. The assessment will be carried out blind by 1 examiner, trained in CRM (Crisis Resource Management) analysis in simulation and debriefing.
Other: Questionnaires — Quality of lige questionnaire Pro-QOL, Karasek questionnaire, Satisfaction questionnaire at work : WRQoL, Work Life Balance scale, Mayo Hight Team Performance scale will be completed at baseline and at 6 months

SUMMARY:
The lack of specific, personalized training for intensive care workers can lead to a deterioration in quality of life at work, and can result in burnout, absenteeism or wanting to leave the service. The aim of this study is to assess the impact of in situ simulation on quality of work life and the effectiveness of multi-professional teamwork in intensive care.

DETAILED DESCRIPTION:
Paramedics in intensive care are particularly exposed to the risk of burnout, which is multifactorial (psychologically and physically challenging environment, life-threatening emergency context, etc.). Personal assistance professions require a high level of compassion, leading to a positive feeling of compassionate satisfaction, i.e. the satisfaction of helping others. Compassion fatigue leads to a reduction in job satisfaction, culminating in burnout. Factors negatively influencing compassion satisfaction are the absence of specific and adapted training, or the lack of support from the hierarchy. Among the pedagogical tools available, in situ simulation could be used to respond to a specific and personalized training request from a care department. The study will be carried out in the cardio-thoracic intensive care unit at Montpellier University Hospital, comparing 2 groups to assess the effect of simulation on paramedics. Paramedics will be randomized into 2 groups, with stratification on diploma (nursing assistant or nurse): group A benefiting from a simulation program, and group B not benefiting from it during the study.

ELIGIBILITY:
Inclusion Criteria:

* Paramedical staff (nurse and nursing assistant) in the cardiothoracic intensive care unit at Montpellier University Hospital.
* Acceptance of being filmed for direct video transcription during the intervention

Exclusion Criteria:

* Refusal of consent or inability to give consent (guardianship, curatorship)
* Paramedics intending to leave the department before the end of the study.
* Not affiliated to a French social security scheme or not a beneficiary of such a scheme

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Subscale of compassion satisfaction of ProQOL-5 (Professional Quality of Life Scale version 5 | From baseline to the end of the follow up at 6 months
  The ProQOL is composed of 30 questions with 3 subscales : compassion satisfaction, burnout and vicarious trauma. Each response are scored from 1 to 5 . The subscale Compassion Satisfaction is composed of 10 questions. A score ≤ 22 indicates a deterioration in compassion satisfaction.

SECONDARY OUTCOMES:
Burnout subscale of ProQOL-5 | From baseline to the end of the follow up at 6 months
  The ProQOL is composed of 30 questions with 3 subscales : compassion satisfaction, burnout and vicarious trauma. Each response are scored from 1 to 5 . The subscale Burnout is composed of 10 questions. A score ≥42 indicates a hight burnout level
Vicarious trauma subscale of ProQOL | From baseline to the end of the follow up at 6 months
  The ProQOL is composed of 30 questions with 3 subscales : compassion satisfaction, burnout and vicarious trauma. Each response are scored from 1 to 5 . The subscale " Vicarious Trauma " is composed of 10 questions. A score ≥42 indicates a hight vicarious trauma level
Karasek | From baseline to the end of the follow up at 6 months
  The Karasek self-questionnaire assess the "job strain ". It is composed of 3 susbscales : the psychological demand, the Decision latitude and the Social support at work. A decision-making latitude score < 72 and a Psychological Demand score ≥ 21 is associated with a Job Strain
WRQoL (QwOL) | From baseline to the end of the follow up at 6 months
  The Work-related Quality of Life is composed of 23 questions. It evaluates 6 dimensions: the feeling of being involved in decisions (3 assertions), appreciation of work organization and general satisfaction (7), help with external demands (3), satisfaction with working conditions (3), satisfaction with the ability to do one's job (6) and stress at work (2). A higher score is associated to a highter quality of life at work.
Work-Life Balance scale questionnaire | From baseline to the end of the follow up at 6 months
  The Work-Life Balance scale assess the impact of work on personal quality of life. It is composed of 3 subscales about : Work interferes with personal life (WIPL), Personal interferes with work (PLIW), Satisfaction with quality of personal and work life (WPLE). A high score is associated with significant interference of work with private life
Mayo High Performance Team Scale | From baseline to the end of the follow up at 6 months
  The Mayo High Performance Team Scale is a standardized evaluation scale, designed to meet non-technical teaching objectives named CRM (Crisis Resource Management). This scale assess the effectiveness and performance of teams of emergency care workers
Adverse event | From baseline to the end of the follow up at 6 months
  Occurrence of adverse events or errors linked to a lack of interprofessional communication

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Departement of anesthesia cardio-thoracic and vascular resuscitation Arnaud de Vinelleuve Hospital CHU of Montpellier., Montpellier, Occitanie
  - University Hospital of Montpellier, Montpellier

IPD SHARING:
Plan to Share IPD: No